CLINICAL TRIAL: NCT04398394
Title: Single Centre Study: Investigational Medical Device of Transscleral Optical Phase Imaging for Retinal Imaging in Healthy Eyes and Retinal Pathology.
Brief Title: Retinal Imaging With Oblique Illumination
Acronym: ASSESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moser Christophe (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Eye Hospital Jules Gonin (Other)
Responsible Party: Sponsor-Investigator, Moser Christophe, Professor, Ecole Polytechnique Fédérale de Lausanne
Organization: Ecole Polytechnique Fédérale de Lausanne (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-00429
Record Dates: First submitted 2020-05-14; First posted 2020-05-21 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Retinal Disease
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Intervention Model Description: Group 1: 20 to 30 individuals with healthy retina, 18 to 50 years old. Group 2: 20 to 30 individuals with healthy retina and presenting with myopia, 18 to 50 years old.
  Group 3: 20 to 30 individuals with healthy retina, over the age of 50. Group 4: 25 to 50 patients with early and intermediate AMD, over the age of 50. Group 5: 25 to 50 patients with other retinopathies than AMD, over the age of 18.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1 (Experimental): Individuals with healthy retina, 18 to 50 years old.
  Interventions: Device: Cellularis version 1 imaging
- Group 2 (Experimental): Individuals with healthy retina and presenting with myopia, 18 to 50 years old.
  Interventions: Device: Cellularis version 1 imaging
- Group 3 (Experimental): Individuals with healthy retina, over the age of 50.
  Interventions: Device: Cellularis version 1 imaging
- Group 4 (Experimental): Patients with early and intermediate AMD, over the age of 50.
  Interventions: Device: Cellularis version 1 imaging
- Group 5 (Experimental): Patients with other retinopathies than AMD, over the age of 18.
  Interventions: Device: Cellularis version 1 imaging

INTERVENTIONS:
Device: Cellularis version 1 imaging — Using a new modality for retinal cell imaging, we aim at comparing qualitatively and quantitatively, the morphology of the deepest layer of the retina, the retinal pigment epithelium (RPE) by imaging the people with a prototype instrument (Cellularis version 1).

SUMMARY:
Retinal diseases are the major cause of blindness in industrialized countries and while tremendous effort is made to develop novel therapeutic strategies to rescue retinal cells, optimal means to evaluate the effects of such treatments is still missing. Nowadays, diseases diagnosis and treatment monitoring are performed thanks to imaging devices and functional measurements (visual acuity of visual field tests). These eye examinations lead to the detection of large scale damages of the retinal tissue, i.e. the diagnosis is made too late or the treatments cannot be adapted in time. With the developed technology, the goal is to provide a tool to the ophthalmologists that allow for better treatment monitoring and early diagnosis. Indeed, the technology is able to image the retinal tissues with a ten times more detailed visualization as compared to the standard of care (OCT instruments, SLO instruments or eye fundus cameras). Towards this goal, we designed the present protocol in order to test the technology with a clinical prototype (Cellularis version 1) in a clinical environment. The objective is to describe and quantify at the cellular level the retina of patient affected by different retinal diseases as well as the healthy retina of people with different ages. We will assess the repeatability of the instrument and compare the results of the measurements with images obtained with the standard of care (OCT and SLO images).

ELIGIBILITY:
Inclusion Criteria:

Group 1

* Individuals, 18 to 50 yo, with normal eye fundus.
* Emmetropic or ametropic between +3D and -3D

Group 2

* Individuals, 18 to 50 yo, with normal eye fundus.
* Myopic between -6D and -12D.

Group 3

* Individuals over the age of 50 and age-matched to patients with AMD.
* With nwith normal eye fundus.
* Astigmatic, myopic (<-12D) or presbyopic participants may be included

Group 4

* Patient over 50 yo, with early or intermediate AMD, including extrafoveolar geographic atrophy
* with visual acuity ≥ 0.6 and clinical judgment of good central fixation.

Group 5

* Patient over 18, with other retinopathy than AMD,
* with visual acuity ≥ 0.6 and nd clinical judgment of good fixation

Exclusion Criteria:

Eye with

* RPE detachment
* a clinically unclear situation
* abnormality preventing good visualization of the fundus
* less than 3 months post-surgery of the anterior segment
* less than 6 months post-surgery of the posterior segment
* active uveitis - myopia ≥12D, hyperopia > +5D, astigmatism > 4D
* contraindication to dilatation
* a palpebral opening that is less than 6 mm in height

Individual:

* albino - unable to fix a target at least 10 seconds
* who does not tolerate being in the dark for 30 minutes
* unable to follow the procedures of the study
* refusing to be informed of the incidental discovery of a clinically significant pathology Investigators of the study, their family members, collaborators and students

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Number RPE [#/mm2] | 2 months
  The primary outcome is the RPE cells density map of the imaged regions (in #/mm2).
Qualitative analysis [unitless] | 2 months
  Together with the quantitative outcomes of the density, a detailed qualitative analysis will also be performed.

SECONDARY OUTCOMES:
averaged RPE cell area [um2] | 2 months
  - The RPE cell area.
Averaged number of neighbors of RPE cells [unitless] | 2 months
  Averaged number of neighbors of RPE cells
Averaged RPE spacing [um] | 2 months
  The averaged RPE spacing in um.
Averaged RPE pigmentation parameter [unitless] | 2 months
  RPE pigmentation parameter at cellular level

CONTACTS AND LOCATIONS:
Overall Officials: Irmela Mantel, MD, Principal Investigator — Jules Gonin eye hospital
Locations (1):
- Jules Gonin eye hospital, Lausanne, Switzerland

REFERENCES:
- [Result] Kowalczuk L, Dornier R, Kunzi M, Iskandar A, Misutkova Z, Gryczka A, Navarro A, Jeunet F, Mantel I, Behar-Cohen F, Laforest T, Moser C. In Vivo Retinal Pigment Epithelium Imaging using Transscleral Optical Imaging in Healthy Eyes. Ophthalmol Sci. 2022 Oct 19;3(1):100234. doi: 10.1016/j.xops.2022.100234. eCollection 2023 Mar. PMID 36545259
- [Derived] Kowalczuk L, Dornier R, Navarro A, Jeunet F, Moser C, Behar-Cohen F, Mantel I. Adaptive Optics-Transscleral Flood Illumination Imaging of Retinal Pigment Epithelium in Dry Age-Related Macular Degeneration. Cells. 2025 Apr 24;14(9):633. doi: 10.3390/cells14090633. PMID 40358157
- See also: Laforest, T., Künzi, M., Kowalczuk, L. et al. Transscleral optical phase imaging of the human retina. Nat. Photonics (2020). — https://doi.org/10.1038/s41566-020-0608-y